CLINICAL TRIAL: NCT05778045
Title: Investigating Patients' Medical Study Experiences in Non-Small Cell Lung Cancer Clinical Trials to Identify Influencing Trends
Brief Title: Examination of Trends in Non-Small Cell Lung Cancer Patients' Medical Study Experiences
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 87324981
Record Dates: First submitted 2023-03-10; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Medical study participation percentages haven't always been fully representative of a given demographic.

The goal is to find out which aspects of a clinical trial may make it more difficult for patients to take part or see it through.

Participating in an observational clinical trial may help patients with non-small cell lung cancer since it advances medical knowledge and may improve treatment choices in the future.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of non-small cell lung cancer
* Patient has self-identified as planning to enroll in a clinical trial for non-small cell lung cancer
* Patient is at least 18 years of age

Exclusion Criteria:

* Inability to perform regular electronic reporting
* Any mental or medical condition that prevents the patient from giving informed consent or participating in the trial
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-small cell lung cancer patients who are actively considering involvement in an observational clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a non-small cell lung cancer clinical study. | 3 months
Number of non-small cell lung cancer patients who remain in clinical trial until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kayser G. [Non-small cell lung cancer. New biomarkers for diagnostics and therapy]. Pathologe. 2015 Nov;36 Suppl 2:189-93. doi: 10.1007/s00292-015-0084-1. German. PMID 26391246
- [Background] Dufraing K, Van Casteren K, Breyne J, D'Haene N, Van Campenhout C, Vander Borght S, Zwaenepoel K, Rouleau E, Schuuring E, von der Thusen J, Dequeker E. Molecular pathology testing for non-small cell lung cancer: an observational study of elements currently present in request forms and result reports and the opinion of different stakeholders. BMC Cancer. 2022 Jul 6;22(1):736. doi: 10.1186/s12885-022-09798-5. PMID 35794532
- [Background] Simeone JC, Nordstrom BL, Patel K, Klein AB. Treatment patterns and overall survival in metastatic non-small-cell lung cancer in a real-world, US setting. Future Oncol. 2019 Oct;15(30):3491-3502. doi: 10.2217/fon-2019-0348. Epub 2019 Sep 9. PMID 31497994

DOCUMENTS (1):
  • Informed Consent Form (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT05778045/ICF_000.pdf